CLINICAL TRIAL: NCT02877277
Title: Restoring Physiological Vitamin C Levels to the Normal Range: Influence on Epigenetic Regulation in Normal and Malignant Hematopoiesis
Brief Title: Epigenetics, Vitamin C and Abnormal Hematopoiesis - Pilot Study
Acronym: EVITA-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Van Andel Research Institute (Other)
Responsible Party: Principal Investigator, Kirsten Grønbæk, Professor, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-16022249
Record Dates: First submitted 2016-08-09; First posted 2016-08-24 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin C (Experimental): Oral intake of vitamin C tablet (500 mg) daily for 56 days
  Interventions: Dietary Supplement: Vitamin C
- Placebo (Placebo Comparator): Oral intake of placebo tablet daily for 56 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Oral intake of vitamin C tablet (500 mg) daily for 56 days
  Arms: Vitamin C
Dietary Supplement: Placebo — Oral intake of placebo tablet daily for 56 days
  Arms: Placebo

SUMMARY:
This study evaluates whether vitamin C improves responses to epigenetic therapy with DNMTis. Half of the patients will receive vitamin C and DNMTi while the other half will receive placebo and DNMTi.

DETAILED DESCRIPTION:
Recently, it was documented that hematological cancer patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) exhibited severe vitamin C deficiency. Vitamin C is an essential co-factor for ten-eleven translocation (TET) enzymes, which initiate DNA demethylation through oxidation of 5-methylcytosine (mC) to 5-hydroxy-methylcytosine (hmC). In-vitro studies show that vitamin C at physiological doses added to DNA methyltransferase inhibitors (DNMTis), induce a synergistic inhibition of cell proliferation and enhanced apoptosis. These effects are mediated via a viral mimicry response recently associated with cancer stem-like cell death and enhanced immune signals including increased expression of bi-directionally transcribed endogenous retrovirus (ERV) transcripts, increased presence of cytosolic double stranded RNAs, and activation of an interferon inducing cellular response to these transcripts. Data suggest that correction of vitamin C deficiency may improve responses to epigenetic therapy with DNMTis. In the EVITA pilot study, the investigators include MDS/AML patients and explore the potential role of restoring vitamin C within the normal physiological range in treatment of hematological cancer with DNMTis.

ELIGIBILITY:
Inclusion Criteria:

* MDS/AML patient in treatment with DNMTi

Exclusion Criteria:

* Intake of vitamin C as a dietary supplement including multivitamin
* Non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-05-29 (Actual)

PRIMARY OUTCOMES:
Overall 5-hmC/5-mC ratio | Change from baseline to day 84
Overall lysine methylation levels | Change from baseline to day 84
5-hmC/5-mC ratio at regulatory genomic regions of genes involved in hematopoietic development | Change from baseline to day 84
Accumulation of 5-hmC/5-mC at regulatory regions of ERVs | Change from baseline to day 84
Aberrant histone methylation associated with hematopoietic development | Change from baseline to day 84
Aberrant histone methylation associated with ERVs | Change from baseline to day 84
Expression levels of ERVs | Change from baseline to day 84
Activity of the viral defense pathway measured by RNA and protein expression | Change from baseline to day 84
ERV specific T-cell recognition in vivo | Change from baseline to day 84

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Grønbæk, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, København Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillberg L, Orskov AD, Nasif A, Ohtani H, Madaj Z, Hansen JW, Rapin N, Mogensen JB, Liu M, Dufva IH, Lykkesfeldt J, Hajkova P, Jones PA, Gronbaek K. Oral vitamin C supplementation to patients with myeloid cancer on azacitidine treatment: Normalization of plasma vitamin C induces epigenetic changes. Clin Epigenetics. 2019 Oct 17;11(1):143. doi: 10.1186/s13148-019-0739-5. PMID 31623675